CLINICAL TRIAL: NCT05037721
Title: Oral Health Initiative With Green Tea,Gargling,Oral Health for Stroke Patients
Brief Title: Effects of Gargling With Green Tea on Oral Health of Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2021-01-021BC
Record Dates: First submitted 2021-08-04; First posted 2021-09-08 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Oral Health
Keywords: green tea; gargling; oral health; stroke patients
MeSH Terms: interventions — Tea; Water

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- gargling with green tea of stroke patients (Experimental): Use fresh green tea (package date less than one month) sourced from the local market and serve in the form of soaked tea bags. 0.5% green tea refers to a tea bag soaked in 0.5g green tea, soaked in 100ml warm water for 5 minutes and let cool. Then, put each bottle of 15ml mouthwash into a disposable opaque bottle, and give two bottles of mouthwash required daily at one time. Use 15ml twice a day, 30 minutes after breakfast and 30 minutes after lunch, each time for 30 seconds. Rinse mouth up and down for 30 seconds. Rinse mouth up and down, half sitting and lying down, and shake the head of bed for 30 degrees. After breakfast, the experimental group and the control group were instructed to clean their teeth according to routine procedures, and telephone reminders were provided to inform them to gargle.
  Interventions: Other: gargling with green tea
- gargling with water of stroke patients (Active Comparator): Use water 15ml of mouthwash into a disposable opaque bottle, and give two bottles of mouthwash required daily at one time. Use 15ml twice a day, 30 minutes after breakfast and 30 minutes after lunch, each time for 30 seconds. Rinse mouth up and down for 30 seconds. Rinse mouth up and down, half sitting and lying down, and shake the head of bed for 30 degrees. After breakfast, the experimental group and the control group were instructed to clean their teeth according to routine procedures, and telephone reminders were provided to inform them to gargle.
  Interventions: Other: gargling with water

INTERVENTIONS:
Other: gargling with green tea — experimental group using 0.5% green tea gargle, control group use clear water gargle, secondary in daily use mouthwash after breakfast and lunch after 30 minutes, 15 ml each use gargle for 30 seconds, total 7 days
  Arms: gargling with green tea of stroke patients
Other: gargling with water — using water gargle, control group use clear water gargle, secondary in daily use mouthwash after breakfast and lunch after 30 minutes, 15 ml each use gargle for 30 seconds, total 7 days
  Arms: gargling with water of stroke patients

SUMMARY:
1. Compare the effects of gargling with green tea on the oral health of stroke patients?
2. Compare whether gargling with green tea can reduce halitosis in stroke patients?
3. Compare whether gargling with green tea can reduce plaque index in stroke patients?

DETAILED DESCRIPTION:
Before the intervention of green tea mouthwash, patients in the experimental group and the control group were tested for oral health status, bad breath and plaque degree, and received routine brushing guidelines. Patients in the experimental group received green tea mouthwash intervention twice a day for 7 day

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients over 20 years of age with acute cerebral stroke admitted by medical institutions.
* Stroke patients diagnosed by medical institutions were treated with the National Institute of Health Stroke Scale; NIHSS) score is 5-15, which is a moderate degree of stroke
* Able to perform mouthwash.
* Those who have passed the three-stage swallowing function screening.
* Those with stable medical condition.

Exclusion Criteria:

* Those who of medical institutes in the diagnosis of severe alzheimer.(ICD-10 code： G30.9)
* Those who severe mental retardation.
* Those has a history of mental illness.
* Those has unable to clearly express their wishes.
* Those has full mouth teeth less than six.
* Those has in the past more than a month use mouthwash.
* Those has treatment of the patients with gingivitis and periodontal disease, oral antibiotics or anti-fungal drugs.
* Those has unable to cooperate or applicable except of assessment tools.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2021-07-30 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
The participants assess the patient's oral health status by the oral health assessment tool scale. | to evaluate the seventh day after use green tea gargle
  Oral Health Assessment Tool (OHAT) kayser-Jones et al. (1995) Oral Health of elderly and cognitively impaired persons. A Brief Oral Health 6 Status Examination was developed. BOHSE) and may be evaluated by a nursing practitioner. Chalmers, Johnson, Tang and Titler developed the Oral Health Assessment Tool (OHAT) after modifying the Simple Oral Health Status Measurement Scale in 2004. This scale can be extended to assess the oral health of elderly people with daily living function dependence, and can be assisted by clinical nursing staff after guidance. The contents of the questionnaire were divided into eight items, including lips, tongue, gums, toothache, saliva, teeth, dentures and oral hygiene. The degree of oral health was divided by 0, 1 and 2 points for each item. The total score ranged from 0 to 16, the higher the score was, the worse the oral health was.

SECONDARY OUTCOMES:
The participants assess the patient's degree of halitosis by the portable breath meter. | to evaluate the seventh day after use green tea gargle
  In this study, a portable breath meter (HC-150®, Tanita Co, Tokyo, Japan) was used to measure the concentration of volatile sulfide in the mouth of patients with a score ranging from 0 to 5. The higher the score, the more severe the halitosis. Manner to ensure that the portable measuring instrument measured the stability of the data, before the study, to perform 20 minutes five patients repeated measurement mouth sulfide values, the research process are made by same nurses within non-executive care plan for all the object of study manner using a portable measuring instrument for testing, in order to maintain consistency measurement. The portable breath meter is calibrated by the instrument to determine the accuracy of the measured value.
The participants assess the patient's the degree of dental plaque with the modified plaque index of "Turesky". | to evaluate the seventh day after use green tea gargle
  In 1962, quigley-Hein developed a plaque index score of 0 to 5 and stained with plaque stains. In 1970, Turesky et al. improved the method. After staining with plaque stains, they scored according to the stained area. The scoring criteria were as follows: 0 was for plaque free; 1. There are scattered punctate dental plaque at the gingival margin of the tooth neck; 2: the width of dental plaque in the neck is less than 1mm(continuous); 3: dental plaque covering area of the tooth neck is more than 1mm, less than 1/3 of the tooth face; 4: the area covered by dental plaque is between 1/3 and 2/3 of the teeth; 5. The dental plaque covers more than 2/3 of the teeth. To distinguish the degree of dental plaque, the total score is 2 points. When the index is greater than 2, it is high; when the index is between 0 and 1, it is low. The higher the score is, the worse the oral health is.

CONTACTS AND LOCATIONS:
Overall Officials: Li ya-wen, Study Director — member
Locations (1):
- Li ya-wen, Taipei, Beitou District, Taiwan

IPD SHARING:
Plan to Share IPD: No